CLINICAL TRIAL: NCT04182321
Title: Metformin as Add-on to the Standard Therapy in Patients With Chronic Hepatitis B: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Metformin as Add-on to the Standard Therapy in Patients With Chronic Hepatitis B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu-Sheng Wang (Other)
Collaborators: Jinan Military General Hospital (Other)
Responsible Party: Sponsor-Investigator, Fu-Sheng Wang, Study Chair, Beijing 302 Hospital
Organization: Beijing 302 Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 960-2019-84
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Chronic Hepatitis B
Keywords: Metformin; Entecavir; chronic hepatitis B; hepatitis B virus
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Metformin; entecavir; Combined Modality Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Therapy (Experimental): Metformin as add-on to entecavir therapy in patients with chronic hepatitis B
  Interventions: Drug: Metformin & Entecavir
- Standard Therapy (Placebo Comparator): Entecavir monotherapy in patients with chronic hepatitis B
  Interventions: Drug: Placebo & Entecavir

INTERVENTIONS:
Drug: Metformin & Entecavir — Adding sustained-release metformin hydrochloride (1000 mg, oral, once a day) for 24 weeks to the ongoing entecavir therapy (0.5 mg, oral, once a day)
  Other Names: Combination Therapy
  Arms: Combination Therapy
Drug: Placebo & Entecavir — Adding placebo (oral, once a day) for 24 weeks to the ongoing entecavir therapy (0.5 mg, oral, once a day)
  Other Names: Standard Therapy
  Arms: Standard Therapy

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial to assess the efficacy and safety of metformin as add-on to entecavir therapy in patients with chronic hepatitis B.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial to assess the efficacy and safety of metformin as add-on to entecavir therapy in patients with chronic hepatitis B. Patients with chronic hepatitis B who met eligibility criteria were randomly assigned (1:1) to receive either metformin (1000 mg, oral, once a day) or placebo (oral, once a day) for 24 weeks in addition to their ongoing entecavir therapy. Patients and investigators were both blinded to group allocation. The primary outcome, serum HBsAg level (log IU/mL) at weeks 24 and 36, was analysed using a linear mixed-effect model. The intention-to-treat populations were included in primary and safety analyses.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg-negative chronic hepatitis B
* Ongoing treatment with Entecavir for more than 12 months
* HBV DNA < 500 IU/mL
* Quantitative HBsAg < 3 log IU/mL
* ALT and AST < 2 × upper limit of normal (ULN)
* Agree to take contraceptive measures during participation for women of a fertile age
* Agree not to engage in other clinical trials during participation
* Understand and sign the informed consent form before taking any steps related to this study

Exclusion Criteria:

* Diabetes mellitus
* Alcoholic liver disease
* Drug-induced liver damage
* Autoimmune liver disease
* Decompensated cirrhosis
* Liver cancer
* Liver transplantation
* Pregnant or lactating women
* Other conditions unsuitable for participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
serum HBsAg level | weeks 24 and 36 after adding metformin or a placebo
  log IU/mL

SECONDARY OUTCOMES:
weight | weeks 24 and 36 after adding metformin or a placebo
  kg
body mass index | weeks 24 and 36 after adding metformin or a placebo
  kg/m^2
fasting glucose | weeks 24 and 36 after adding metformin or a placebo
  mmol/L
HbA1c | weeks 24 and 36 after adding metformin or a placebo
  percentage (%)
triglycerides | weeks 24 and 36 after adding metformin or a placebo
  mmol/L
total cholesterol | weeks 24 and 36 after adding metformin or a placebo
  mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Study Chair — The Fifth Medical Center of Chinese PLA General Hospital (Beijing 302 Hospital)
Locations (1):
- The 960th Hospital of Chinese PLA Joint Logistics Support Force (Jinan Military General Hospital), Tai’an, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data and full study protocol are available upon reasonable request. Researchers should send it to fswang302@163.com to gain access.
Supporting Information: Study Protocol
Time Frame: After publication of the study results
Access Criteria: Researchers interested in our study

REFERENCES:
- [Background] Polaris Observatory Collaborators. Global prevalence, treatment, and prevention of hepatitis B virus infection in 2016: a modelling study. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):383-403. doi: 10.1016/S2468-1253(18)30056-6. Epub 2018 Mar 27. PMID 29599078
- [Background] GBD 2017 Causes of Death Collaborators. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1736-1788. doi: 10.1016/S0140-6736(18)32203-7. Epub 2018 Nov 8. PMID 30496103
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] Xun YH, Zhang YJ, Pan QC, Mao RC, Qin YL, Liu HY, Zhang YM, Yu YS, Tang ZH, Lu MJ, Zang GQ, Zhang JM. Metformin inhibits hepatitis B virus protein production and replication in human hepatoma cells. J Viral Hepat. 2014 Aug;21(8):597-603. doi: 10.1111/jvh.12187. Epub 2013 Oct 24. PMID 24164660
- [Background] Honda M, Shirasaki T, Terashima T, Kawaguchi K, Nakamura M, Oishi N, Wang X, Shimakami T, Okada H, Arai K, Yamashita T, Sakai Y, Yamashita T, Mizukoshi E, Kaneko S. Hepatitis B Virus (HBV) Core-Related Antigen During Nucleos(t)ide Analog Therapy Is Related to Intra-hepatic HBV Replication and Development of Hepatocellular Carcinoma. J Infect Dis. 2016 Apr 1;213(7):1096-106. doi: 10.1093/infdis/jiv572. Epub 2015 Nov 29. PMID 26621908